CLINICAL TRIAL: NCT06342089
Title: Prevalence And Severity Of Molar Incisor Hypomineralization Among A Group Of Children With Type I Diabetes Milletus:A Cross Sectional Study.
Brief Title: Prevalence And Severity Of Molar Incisor Hypomineralization Among A Group Of Children With Type I Diabetes Milletus.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Samir Fahmy Auob, Resident doctor at the Department of Pediatric Dentistry, Cairo University
Other Study IDs: NCT06342089
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization (MIH); Type I diabetes milletus(TIDM)
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with type I diabetes milletus: •Patient aged 8 to 14 years and diagnosed with type I diabetes milletus with erupted all 4 first permanent molars.
  Interventions: Other: Type I diabetes milletus

INTERVENTIONS:
Other: Type I diabetes milletus — the exposure is type I diabetes milletus

SUMMARY:
* Determine the prevalence of molar incisor hypomineralization among a group of children with type I diabetes millutes, its severity and treatment need via clinical examination of children with type I diabetes millutes .
* Teeth will be cleaned gently using gauze and wet with saliva during examination. A disposable diagnostic set (mirror, probe) will be used for each patient where mirrors will be used for proper visualization especially for maxillary teeth.
* Blunt explorers will be used to aid in tactile sensation if needed, as during the differentiation between rough and smooth enamel edges and/or during the inspection of the caries extent if it exists. No diagnostic radiographs will be taken.
* The severity and treatment needs of each case with MIH will be recorded in patient's chart.
* The results of the study will be regularly monitored by the supervisors who will have full access to these results.

DETAILED DESCRIPTION:
* This cross-sectional study will be carried out by recruiting a sample of participants previously diagnosed with type I diabetes millutes.
* Details regarding participant diagnosis and treatment of type I diabetes millutes will be obtained from medical records. This includes date and the age of the child on diagnosis type I diabetes millutes, and a recent HbA1c level analysis within three months of the dental examination.
* A disposable diagnostic set (mirror, probe) were used for each child to examine the four first permanent molars , the four maxillary ,the four mandibular incisors and second primary molars to detect the presence of molar incisor hypomineralization and its severity and scores will be recorded in the chart then it will be correlated with treatment need.
* The teeth affected with molar incisor hypomineralization will be treated according to the recommendations of European academy of pediatric dentistry and the intervention will be recorded in patient's chart.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 8 to 14 years and diagnosed with types I diabetes milletus.
* Eruption of all 4 first permanent molars.
* Acceptance to participate.

Exclusion Criteria:

* Presence of orthodontic appliance.
* Patient with any other type of enamel defect.
* Patients with any other systemic conditions rather than types I diabetes milletus that may affect tooth development.

Ages: 8 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: * This cross-sectional study will be carried out by recruiting a sample of participants previously diagnosed with types I diabetes milletus aged from( 8-14) accept to participate.
  * All permanent molars must be erupted as the diagnosis of molar incisor hypomineralization required at least one permanent molar involved .
  * The patient mustn't have any other medical conditions nor orthodontic appliance that may affect the enamel quality
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of molar incisor Hypomineralization among among a group of children with type I diabetes milletus. | one year
  The prevalence will be measured according to the diagnostic criteria of molar incisor Hypomineralization established by European Academy of Pediatric Dentistry.
  Measuring unit: percentage

SECONDARY OUTCOMES:
Severity of molar incisor Hypomineralization among among a group of children with type I diabetes milletus. | one year
  the severity will be measured according to:European Academy of Paediatric Dentistry (EAPD) criteria.
  Measuring unit: Categorical
Treatment need | one year
  The treatment need will be measured according to: treatment need index Measuring unit: Categorical l

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cingolani R, Stolz W, Ploog K. Electronic states and optical transitions in modulation-doped n-type GaxIn1-xAs/AlxIn1-xAs multiple quantum wells. Phys Rev B Condens Matter. 1989 Aug 15;40(5):2950-2955. doi: 10.1103/physrevb.40.2950. No abstract available. PMID 9992226
- [Background] Ghanim A, Silva MJ, Elfrink MEC, Lygidakis NA, Marino RJ, Weerheijm KL, Manton DJ. Molar incisor hypomineralisation (MIH) training manual for clinical field surveys and practice. Eur Arch Paediatr Dent. 2017 Aug;18(4):225-242. doi: 10.1007/s40368-017-0293-9. Epub 2017 Jul 18. PMID 28721667
- [Background] Lygidakis NA, Garot E, Somani C, Taylor GD, Rouas P, Wong FSL. Best clinical practice guidance for clinicians dealing with children presenting with molar-incisor-hypomineralisation (MIH): an updated European Academy of Paediatric Dentistry policy document. Eur Arch Paediatr Dent. 2022 Feb;23(1):3-21. doi: 10.1007/s40368-021-00668-5. Epub 2021 Oct 20. PMID 34669177
- [Background] Steffen R, Kramer N, Bekes K. The Wurzburg MIH concept: the MIH treatment need index (MIH TNI) : A new index to assess and plan treatment in patients with molar incisior hypomineralisation (MIH). Eur Arch Paediatr Dent. 2017 Oct;18(5):355-361. doi: 10.1007/s40368-017-0301-0. Epub 2017 Sep 14. PMID 28913739
- [Background] Mast P, Rodrigueztapia MT, Daeniker L, Krejci I. Understanding MIH: definition, epidemiology, differential diagnosis and new treatment guidelines. Eur J Paediatr Dent. 2013 Sep;14(3):204-8. PMID 24295005